CLINICAL TRIAL: NCT03001986
Title: Effectiveness and Safety of Inactivated EV71 Vaccine (Human Diploid Cell) in 6-71 Months Children: an Open-label Controlled Phase Ⅳ Clinical Study
Brief Title: The Phase IVb of Inactivated Enterovirus 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-012-03
Record Dates: First submitted 2016-09-17; First posted 2016-12-23 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Hand, Foot and Mouth Disease (HFMD)
Keywords: effectiveness; safety; hand, foot and mouth disease (HFMD); Enterovirus A, Human; vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vaccine (3.0 EU) (Experimental): healthy children (6-71 months old) have been injected by inactivated EV71 vaccine (KMB-17) of 3.0 EU (neutralization antibodies titer unit; 100 U in phase III clinical trials, or 320 EU (Elisa assay unit) in phase I and II clinical trials)
  Interventions: Biological: inactivated EV71 vaccine (KMB-17 cells)

INTERVENTIONS:
Biological: inactivated EV71 vaccine (KMB-17 cells) — Receiving 2 doses of the EV71 inactivated vaccine at an interval of 1 month.

SUMMARY:
Enterovirus 71 (EV71), a major pathogen causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Its infection occasionally leads to severe diseases and death, with central nervous system (CNS) damage.

An inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been finished phase I, II and III clinical trials and licensed by CFDA in China at Dec. 3, 2015. Based on the results of clinical trials, the protective efficacy of inactivated EV71 vaccine is 97% against HFMD caused by EV71. The target population is determined to be susceptible children aged 6 to 71 months; this target population is well known as a major global population with strict requirements for safety and efficacy of vaccines in implementing the World Health Organization (WHO) Expanded Program on Immunization (EPI) . Thus, it is necessary and significant to conduct a postmarketing phase IV trial in large populations for long-term observation to evaluate the distinctive effectiveness and to identify potential safety issues .

This study is an open-label and controlled postmarketing phase IV trial on children aged 6-71 months who resided in 3 districts of Xiangyang City, Hubei Province, China.

DETAILED DESCRIPTION:
Primary Objective: To evaluate the effectiveness of EV71 vaccine after mass vaccination in a large population (Chinese healthy children aged 6-71 months) for preventing against EV71-associated hand, foot and mouth disease.

Secondary Objective: To evaluate the safety of EV71 vaccine after mass vaccination in a large population (Chinese healthy children aged 6-71 months).

Participants: The children aged 6-71 months in the study area registered in August 2016 in the Childhood Immunization Information Management System (CIIMS) in Hubei Province are designated as study population. Of these children, 39189 will be recruited in the vaccine group for receiving 2 doses of EV71 inactivated vaccine at an interval of 1 month. The remaining children will be used as the control group.

Sampling size: The total sample size is primarily calculated based on the previous HFMD monitoring data of the study sites from 2010 to 2015 by stratifying the data into 6 age groups as follows: 6-11 months, 12-23 months, 24-35 months, 36-47 months, 48-59 months and 60-71 months, respectively. Prior to the identification of minimum annual HFMD incidences caused by EV71 infection are 0.08%-6.05% (data not shown). Assuming a vaccine effectiveness of 90% , power of 0.80 with a 0.05 significance level (two-tailed), and drop-out rate of 20% , the sample size would be 39189 in the vaccine group.

Standard Operating Procedures:

1. Recruitment among the study population.
2. Recruit the study participants, and the children's guardians sign the informed consent.
3. The participants receive the 1st dose EV71 vaccine.
4. Observation for 30 minutes after vaccination in the vaccination clinic.
5. Follow up the enrolled participants by using contact card for recording any occurred AEs of for a period of 30 days p.i. through home visits (in villages) or telephone visits (in urban communities) within 30 days p.i. the first injection.
6. The participants receive the 2nd dose EV71 vaccine.
7. Observation for 30 minutes after vaccination in the vaccination clinic.
8. Follow up the enrolled participants by using contact card for recording any occurred AEs of for a period of 30 days p.i. through home visits (in villages) or telephone visits (in urban communities) within 30 days p.i. the second injection.
9. Twenty-eight days p.i.of the 2nd vaccination dose, conduct HFMD case surveillance on all participants in the vaccine and control groups for a follow-up period of up to 14 months through the database of Notifiable Infectious Diseases Network in Hubei, and detect EV71 in associated feces or anal swab specimens that are collected at hospitals or Community Healthcare Service Centers by real-time PCR (RT-PCR).

Statistical Analysis Plan:

Primary statistical analysis will be to calculate the vaccine effectiveness against EV71-associated HFMD, and to compare incidence density of EV71-associated HFMD between vaccine group and control group.

Secondary analyses will be to calculate the vaccine effectiveness against EV71-associated severe HFMD and EV71-associated hospitalized HFMD, and to describe adverse events in the vaccine recipients.

Quality Assurance Plan:

1. Training Investigators: Administrative and technical personnel at all levels in study areas are required to participate in training on the study objectives, enrollment procedures, follow-up requirement, data collection, quality control measures, sample handling and transport, and all other operations involved.
2. Supervision and Monitoring: Institute of Medical Biology, Chinese Academy of Medical Science (IMBCAMS) and the Hubei province Center for Control and Prevention (Hubei CDC ) will supervise and monitor vaccination clinic during the implementation period according to the progress of study; and the Xiangyang City Center for Control and Prevention will supervise and monitor each vaccination clinic on selected appointment days. The focus of supervision and monitoring will be to observe whether the vaccination clinics strictly follow protocols and procedures and any problems found can be quickly resolved with timely feedback. Any serious and consistent problems will be reported to the higher level, so that corrections can be made timely.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (6-71 months old children)
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol

Exclusion Criteria:

* Allergy to a vaccine , any ingredient of vaccine or substance used in the preparation process including excipients, formaldehyde, and kanamycin sulfate.
* Fever, acute illness
* Severe chronic disease, allergic diathesis

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40724 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The effectiveness of inactivated EV71 vaccine in preventing hand-foot-and-mouth disease (HFMD) caused by Enterovirus 71 (EV71) in large scale population of Chinese children (from 6 to 71 months old) in Hubei Province, China. | Up to 14 months from twenty-eight days p.i.of the 2nd vaccination dose
  The effectiveness of inactivated EV71 vaccine and 95% confidence intervals were calculated on the basis of the observed difference of incidence between the children (from 6 to 71 months old) who were vaccinated and those who were not vaccinated.

SECONDARY OUTCOMES:
Incidence of treatment adverse events | Within 30 days postinoculation each dose
  The adverse events were observed and recorded within 30 minutes post immunization (p.i.), within 30 days after the 1st injection, as well as after the 2nd injection.

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Guan, M.S., Principal Investigator — Hubei Province Center for Diseases Control and Prevention
Locations (1):
- Hubei Province Center for Diseases Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Participants do not agree to share individual data.

REFERENCES:
- [Derived] Guan X, Che Y, Wei S, Li S, Zhao Z, Tong Y, Wang L, Gong W, Zhang Y, Zhao Y, Wu Y, Wang S, Jiang R, Huang J, Liu Y, Luo W, Liao Y, Hu X, Zhang W, Dai Y, Jiang G, Min G, Liu F, You X, Xu X, Li J, Li C, Fan S, Hang L, Huang Q, Li Q. Effectiveness and Safety of an Inactivated Enterovirus 71 Vaccine in Children Aged 6-71 Months in a Phase IV Study. Clin Infect Dis. 2020 Dec 3;71(9):2421-2427. doi: 10.1093/cid/ciz1114. PMID 31734699